CLINICAL TRIAL: NCT06437106
Title: The Effect of Maternally Scent-digested Blanket on the Stress Level, Crying Duration and Physiological Parameters of Premature Newborns
Brief Title: The Effect of Maternally Scent-digested Blanket on Stress, Crying and Physiological Parameters of Premature Newborns
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Shahla Shafaati Laleh, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SSL&APM
Record Dates: First submitted 2024-04-09; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Family-centered Care
Keywords: The smell of mother; baby; stress; physiological parameters
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Intervention group one includes premature babies who receive a blanket impregnated with the mother's smell.
  The second intervention group includes premature babies who receive a blanket without the smell of the mother.
  The control group includes premature babies who do not receive any intervention and receive routine care.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A blanket impregnated with the mother's odor (Active Comparator): Intervention group 1 consists of premature babies who receive a blanket impregnated with the mother's odor.
  Interventions: Behavioral: A blanket impregnated with the mother's odor
- blanket without mother's smell (Active Comparator): Intervention group 2 includes premature babies who receive a blanket without the smell of the mother.
  Interventions: Behavioral: blanket without mother's smell
- control group (Active Comparator): The control group includes premature babies who receive no intervention and receive routine care.
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: A blanket impregnated with the mother's odor — Intervention group 1 consists of premature babies who receive a blanket impregnated with the mother's odor.
  Arms: A blanket impregnated with the mother's odor
Behavioral: blanket without mother's smell — Intervention group two consists of preterm infants who receive blanket without mother's odor.
  Arms: blanket without mother's smell
Behavioral: control group — The control group includes premature babies who are not subjected to any intervention and receive the usual care.
  Arms: control group

SUMMARY:
Olfaction is a highly developed and crucial sensory modality that connects the infant and the mother, facilitating the infant's ability to locate and reach the mother's breast. the olfactory important sensory ability develops during intrauterine life . By the 11th week of pregnancy, human embryos have completely developed olfactory cells, indicating the complete formation and functionality of the olfactory sensory system during the first trimester . Hence, the olfactory sense undergoes development between the 26th and 28th weeks of pregnancy and, like other senses, plays a role in producing both motor and emotional responses .The mature olfactory system of newborn infants also effectively reduces pain and distress. The results of some studies have shown that the mother's voice and the smell of breast milk can reduce discomfort scores and analgesic effects during painful procedures . Odors can trigger the release of neurotransmitters, such as endorphins, in infants. Neurotransmitters are released in infants to alleviate painful stimuli, leading to a drop in stress levels . Researchers clinical experience shows that covering the baby calms and reduces crying. But no evidence-based studies have been conducted.

The present study is planned in the form of a randomized controlled trial design and will investigate the effect of a blanket impregnated with the mother's scent on the amount of stress, duration of crying and physiological parameters of premature infants admitted to the NICU.

Hypotheses:

In premature newborns;

H1: Covering with a blanket with maternal scent digested reduces the stress level of newborns.

H2: Covering with a blanket with maternal scent digested reduces the crying time of newborns.

H3: Covering with a blanket with maternal scent digested positively affects the physiological parameters of newborns.

H4: Covering with a blanket with maternal scent digested is more effective in reducing the stress level of newborns than covering with a blanket without maternal scent and the control group (babies not covered).

H5: Covering with a blanket with maternal scent digested is more effective in reducing the crying time of newborns than covering with a blanket without maternal scent and the control group (babies not covered).

H6: Covering with a blanket with maternal scent digested affects the physiological parameters of newborns more positively than the cover with maternal scent undigested and the control group (babies not covered).

DETAILED DESCRIPTION:
When preterm babies are admitted to the NICU, preterm babies are deprived of mother's hugs, sounds, and smells. Maternal involvement has recently been recognized as an important aspect of the care of hospitalized preterm infants that has a positive impact on clinical outcomes. Standard care in babies can cause stress, and following may cause pain in the baby over time. Both pharmacological and non-pharmacological approaches are used together to alleviate pain and reduce stress in infants. One of the non-medicinal methods is maternal odor. Researches has indicated that maternal odors, including breast milk, body odor, and amniotic fluid, particularly the odor of breast milk, can decrease stress reactions in newborn infants, such as crying and motor activity . The present study will be conducted with the aim of determining the effect of a blanket impregnated with the mother's smell on the amount of stress, crying duration and physiological parameters of premature babies

Method:

Place of the Research :

The data of current study will be collected on premature babies hospitalized in the neonatal intensive care unit of Al-Zahra Teaching and Research Hospital and Taleghani Teaching and Research Hospital, which are mother and baby friendly hospitals in Tabriz city.

Sample research:

TG*Power software (latest ver. 3.1.9.7; Heinrich-Heine Universität Düsseldorf, Düsseldorf, Germany) was used to determine the sample size in the study. In the study, Rad (2021)** investigated the effect of the smell of breast milk and the smell of another mother's breast milk on the behavioral responses to pain caused by hepatitis B (HB) vaccine injection in preterm babies. In the study, a significant difference was observed for peak heart rate values, and intra-group and inter-group differences were calculated. In the smell of breast milk group, the pretest mean heart rate was 139 ± 16.1 points and the posttest mean was 146 ± 14.3 points. In the another mother's breast milk group, the pretest mean heart rate was 141 ± 15.6 points and the posttest mean was 153 ± 15.5 points. In the control group, the pre-test average heart rate was 139 ± 17.8 points and the post-test average was 155 ± 17.7 points. Power was calculated using the "ANOVA: Repeated measures, within-between interaction" method for two repeated measurements of heart rate averages in three groups. As a result, was determined that should be 54 observations in the sample with a statistical power level of 80% and a significance level of 5% for the calculated (f=0.220)* effect size. Considering sample loss (10%) such as dropping out of the study, will be sufficient to work with at least 60 participants. Participants will be grouped with 20 participant in each group.

Data collection tools: Mother and baby information form, baby monitor which is used to evaluate the baby's heart rate and oxygen saturation level and the baby's temperature, , stopwatches designed to count the baby's breathing and crying time, baby stress scale and evaluation form Babies will be used.

Application of the research:

Before the start of data collection, the family of an infant who meets the selection criteria planned for the research is informed about the purpose and content of the research, and they are asked if they want to participate in the study and their written consent is obtained. Through the "informed consent form". Before conducting, the research will be explained to midwives, doctors and other personnel working in the research unit. Necessary tools will be available before conducting (stopwatch, blanket,...). In this research, random allocation will be done through random blocks with the size of blocks of 6 and 9 and with the allocation ratio of 1:1:1. In order to hide the allocation of the type of intervention, it will be written on a sheet of paper and placed inside the opaque envelopes and numbered consecutively. The envelopes will be determined according to the order of the participants entering the open study and the type of intervention received. Random allocation and allocation concealment will be done by a person not involved in sampling and data collection. A square shaped blanket (made of cotton fabric) is given to the mother for one night, as in Jessen's (2020) study, placed in contact with and between the breasts of the showered mother, so that the blanket is impregnated with the mother's scent. to be The mother is asked to keep the blanket in the sealed plastic bag given to her during the day and to use her regular shampoo, regular soap. and avoid using new products. All blankets are washed with the same detergent before giving to the mother. Babies covered with a blanket impregnated with their mother's scent formed group 1 (20 participant), babies covered with a blanket not covered with their mother's scent, group 2 (n = 20) and babies in the control group, which was not covered with any blanket. , forms group 3 (20 participant). All babies' diapers are changed and cleaned at least half an hour before the operation. Babies will be fed. In order to prevent heat loss and create equal conditions, this method is performed with a naked baby (with diapers) in the incubator. No painful procedures will be performed on the day of the request, at least half an hour before and half an hour after. Before the intervention, i.e. 5 minutes before the measurement (blanket impregnated with mother's smell and plain blanket without mother's smell), the premature baby is evaluated and the stress level and physiological parameters are observed and recorded. This process starts for one hour in the morning. Observation by the researcher from before the intervention to after the intervention to evaluate the stress level, duration of crying and physiological parameters of the babies is taken 5 minutes before the intervention, immediately after the intervention, every 15 minutes during the intervention and 5 minutes after the intervention. . . The stress level is evaluated by observation by the researcher who does not know which group the babies are in. In addition, the infant's physiological parameters are evaluated 5 minutes before the intervention, immediately after the intervention, every 15 minutes during the intervention and 5 minutes after the intervention by the same researcher. During the intervention, the baby will be left alone to avoid affecting stress symptoms, crying duration and physiological parameters, and 30 minutes after the procedures performed on the baby, the intervention will take place and no other actions will be performed during the intervention.

intervention group; Blanket group impregnated with mother's smell: (intervention group 1)

1. Parents of babies in intervention group 1 first fill out the "Mother and Baby Information Form".
2. A blanket impregnated with the smell of the mother is covered over the baby for one hour in the morning for three days.
3. The stress level of babies is evaluated by the researcher through observation before, during and after the intervention.
4. Physiological parameters of babies and duration of crying are evaluated by the same observer.
5. Heart rate and oxygen saturation of the baby are checked and recorded before, during and after the intervention.
6. When the treatment and care is not done on the baby, the research procedure will be done.

Simple blanket group without mother's smell: (intervention group 2)

1. Parents of babies in intervention group 2 first fill in the "Mother and Baby Information Form".
2. A blanket that does not smell of the mother and is simple is covered over the baby for three days in the morning for one hour.
3. The stress level of babies is evaluated by the researcher through observation before, during and after the intervention.
4. Physiological parameters of babies and duration of crying are evaluated by the same observer.
5. Heart rate and oxygen saturation of the baby are checked and recorded before, during and after the intervention.
6. When the treatment and care is not done on the baby, the research procedure will be done.

control group:

1. Babies in the control group first fill out the "Mother and Baby Information Form".
2. The usual care method of the unit will be applied to the baby without any intervention.
3. The amount of stress of the babies is evaluated by the researcher through observation in the morning at the same time as the babies of the intervention group.
4. Physiological parameters of babies and duration of crying are evaluated by the same observer.
5. The baby's heart rate and oxygen saturation are checked and recorded.
6. When the treatment and care is not done on the baby, the research procedure will be done

Research data analysis:

The data obtained in the research will be analyzed using SPSS software for Windows 24.0. In data evaluation, number, percentage, average and standard deviation will be used as descriptive statistical methods. Before conducting the hypothesis tests, data distribution characteristics are checked with the Kolmogorov Smirnov test, skewness and homogeneity of variance are checked with Levene's test, and if conditions exist, the independent sample t test is checked. T test is used to compare continuous data between two independent groups. Otherwise, the Mann Whitney U test is used to compare continuous data between more than two independent groups. One-way Anova test will be used for comparison, if not available, Kruskal Wallis tests will be used. After one-way ANOVA test, Benforrini and Tukey tests will be used as additional post-hoc analysis to determine differences. And two-by-two Mann Whitney U tests are used for the Kruskal Wallis test. Among the continuous variables of the research, the correlation analysis will be evaluated and the classified data will be evaluated with the chi-square test. In all analyses, values of p<0.05 (two-sided) will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* The baby is in the neonatal period (babies between 0 and 28 days),
* Admission to the neonatal intensive care unit has been completed.
* Between 28 and 36 weeks of pregnancy,
* The general situation is stable.
* Not having conditions that prevent pain assessment (intracranial bleeding, neuromotor development delay, etc.),
* The child has not been sedated or sedated in the last 6 hours.
* Baby's breastfeeding should be finished 30 minutes before the intervention. Its weight is more than 1000 grams.
* Apgar score is high,
* Consent of the families to participate in the research

Exclusion Criteria:

Hospitalized for a second time during the data collection process. Lack of literacy in parents

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Infant stress level: | The stress level of the baby will be evaluated 5 minutes before the intervention, immediately after the intervention, every 15 minutes during the intervention and 5 minutes after the intervention for a total of one hour for 3 consecutive days.
  The stess levels of the infants will be evaluated via Infant stress scale. Infant stress scale was developed by Ceylan and Bolışık for assessing stress in premature infants contains 24 items: "facial expression", "body color", "breathing", "activity level", "relaxation", "muscle tone". ", "end limbs" and "body posture" consists of 8 subgroups: it is enough for the baby to show only one of the behaviors in each of the items for scoring. If the baby shows both signs (behavior) in Each of the items in the table (for example, both scores 1 and 2 will be the highest score for the action. This scale is designed on a 3-point Likert scale between 0 and 2 points). The maximum is 16 points and the minimum is 0 points. The higher the stress score, the higher the stress level of the baby is evaluated by the researcher.
Oxygen saturation measurement: | Oxygen saturation of the baby will be measured 5 minutes before the intervention, immediately after the intervention, every 15 minutes during the intervention and 5 minutes after the intervention, for a total of one hour for 3 consecutive days.
  The oxygen saturation levels of the baby will be measured by a monitor that is connected to the baby and shows the level of oxygen saturation. The observation is done by the researcher.
Respiratory rate/minute: | The infant's breathing is measured 5 minutes before the intervention, immediately after the intervention, every 15 minutes during the intervention and 5 minutes after the intervention, for a total of one hour for 3 consecutive days.
  A stopwatch will be use to determine the respiratory rate in a minute of babies. The evaluation is done by the researcher.
Body temperature: | The baby's temperature is measured 5 minutes before the intervention, immediately after the intervention, every 15 minutes during the intervention and 5 minutes after the intervention, for a total of one hour for 3 consecutive days.
  Through a monitor that shows the baby's skin temperature. The temperature is recorded in Celsius in the newborn assessment form. The evaluation is done by the researcher.
Heart rate/minute: | The baby's heart rate will be measured 5 minutes before the intervention, immediately after the intervention, every 15 minutes during the intervention and 5 minutes after the intervention, for a total of one hour for 3 consecutive days.
  To determine the baby's heart rate, a monitor that is connected to the baby and measures the heart rate/minute will be used. The evaluation is done by the researcher.
The duration of the baby's crying: | The duration of the baby's crying is measured for one hour during the evaluation process. This will be done for 3 consecutive days
  A stopwatch will be used to determine the duration of the baby's crying. The evaluation will be done by the researcher. The duration of the baby's crying in seconds will be recorded in the baby's evaluation form

CONTACTS AND LOCATIONS:
Overall Officials: shahla shafaati laleh, Master, Principal Investigator — Turkey , Istanbul University- cerrahpasha
Locations (1):
- Istanbul - cerrahpasha University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No